CLINICAL TRIAL: NCT05991531
Title: Dynamic Changes of Serum HBV RNA in Chronic Hepatitis B Patients With Low Level HBV DNA Treated With Nucleoside (Acid) Analogues
Brief Title: Dynamic Changes of Serum HBV RNA in Chronic Hepatitis B Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Serum HBV RNA
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Chronic Hepatitis B Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Some patients with low-level viremia (LLV) are also likely to develop hepatocellular carcinoma (HCC) or other liver diseases. The relationship between HBV RNA levels and fibrosis in patients with HBV DNA negative or LLV is still lacking evidence. The purpose of this study is to observe the differences in HBV RNA levels and their association with efficacy in HBV DNA negative or LLV patients. Investigators conduct the prospective, single-center, non-randomized, observational clinical study. A total of 100 chronic hepatitis B (CHB) patients who receive antiviral therapy with nucleoside (acid) analogues for 1-3 years will be enrolled. The enrolled patients will be followed up five times to collect clinical data and record adverse events (at baseline, week 12, week 24, week 36 and week 48, respectively).

ELIGIBILITY:
Inclusion Criteria:

* 1.18 years old or above and the gender is not limited;
* 2. Patients who receive antiviral therapy with nucleoside (acid) analogues for 1-3 years ;
* 3. Patients with HBV DNA negative (HBV DNA<20 IU/ml) or LLV（HBV DNA 20-2000 IU/mL）
* 4. Good compliance and voluntary signing of informed consent.

Exclusion Criteria:

* 1. Patients with decompensated cirrhosis;
* 2. Patients co-infection with other viruses, such as hepatitis A virus, hepatitis C virus, hepatitis D virus, hepatitis E virus, HIV virus, etc.;
* 3. Patients with significant renal, cardiovascular, pulmonary, or neurological disease;
* 4. Patients have active or suspected malignancy or history of malignancy;
* 5. Patients who were identified not appropriate for the study by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who receive antiviral therapy with nucleoside (acid) analogues for 1-3 years and with HBV DNA negative or LLV.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The decrease of HBV RNA from baseline to 48 weeks | 2023.8-2025.8
  The investigators detect the dynamic change of HBV RNA and the decline from baseline to 48 weeks;

SECONDARY OUTCOMES:
HBV RNA undetectable rate at 48 weeks; | 2023.8-2025.8
  After 48 weeks of treatment after enrollment, the investigators detect the HBV RNA undetectable rate 48 weeks;
The association of the dynamic changes of serum HBV RNA levels with HBsAg and HBeAg levels; | 2023.8-2025.8
  During 48 weeks of treatment, the investigators detect the association of the dynamic changes of serum HBV RNA levels with HBsAg and HBeAg levels;
The association of HBV RNA changes with the liver stiffness; | 2023.8-2025.8
  During 48 weeks of treatment, the investigators detect the association of HBV RNA changes with the liver stiffness;

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China